CLINICAL TRIAL: NCT03836924
Title: A Prospective, Multicenter, Post-marketing Surveillance to Assess Safety & Efficacy of Perampanel in Indian Patients as An Adjunctive Treatment in Partial Onset Seizures With or Without Secondary Generalized Seizures in Patients With Epilepsy Aged 12 Years or Older
Brief Title: A Study to Assess Safety and Efficacy of Perampanel in Indian Participants as an Adjunctive Treatment in Partial Onset Seizures With or Without Secondary Generalized Seizures in Participants With Epilepsy Aged 12 Years or Older
Status: Completed | Type: Observational
Sponsor: Eisai Pharmaceuticals India Pvt. Ltd (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: E2007-M091-508
Record Dates: First submitted 2019-02-08; First posted 2019-02-11 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Partial Onset Seizures; Epilepsy
Keywords: E2007; Fycompa; Perampanel; Prospective; Partial onset seizures; Epilepsy; Seizures
MeSH Terms: conditions — Epilepsy; Seizures | interventions — perampanel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Perampanel: Participants receiving perampanel tablets, orally according to prescribing information and the treating physician's clinical judgment will be observed prospectively for up to 6 months or participant withdrawal, whichever occurs first.
  Interventions: Drug: Perampanel

INTERVENTIONS:
Drug: Perampanel — Perampanel tablets.
  Other Names: E2007; Fycompa

SUMMARY:
The purpose of this study is to assess the safety of perampanel in the treatment of partial onset seizures in participants of age 12 years and older with epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Participants prescribed perampanel for the adjunctive treatment of partial onset seizures based on independent clinical judgment of treating physicians.

Exclusion Criteria:

* Participation in another study involving administration of an investigational drug or device whilst participating in this observational study.
* Hypersensitivity [allergic] to perampanel.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Indian participants with epilepsy aged 12 years or older.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants Reporting one or More Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Up to 6 months

SECONDARY OUTCOMES:
Percent Change From Baseline in Seizure Frequency per 28 days During the Treatment Period | Up to 6 months
Percentage of Participants Who Experienced at Least 50 Percent Reduction From Baseline in Seizure Frequency During the Treatment Period | Up to 6 months
Percentage of Participants Who Achieved a Seizure-free Status During the Treatment Period | At 3 months and 6 months

CONTACTS AND LOCATIONS:
Locations (12):
- India (12):
  - BGS Gleneagles Global Hospitals, Bengaluru, Karnataka
  - Seth G S Medical College & KEM Hospital, Mumbai, Maharashtra
  - Brain Clinic, Jasleen Hospital, Nagpur, Maharashtra
  - Getwell Hospital and Research Institute, Nagpur, Maharashtra
  - Deenanath Mangeshkar Hospital and Research Centre, Pune, Maharashtra
  - Lifepoint Multispecialty Hospital, Pune, Maharashtra
  - Nizam's Institute of Medical Sciences Department of Neurology, Hyderabad, Telangana
  - Sanjay Gandhi Post Graduate Institute of Medical Sciences, Lucknow, Uttar Pradesh
  - Ramakrishna mission seva pratisthan vivekananda institute of medical sciences, Kolkata, West Bengal
  - Sri Aurobindo Seva Kendra, Kolkata, West Bengal
  - Shri Ganga Ram Hospital, Delhi
  - Advance Neurology & Superspeciality Hospital, Jaipur

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.